CLINICAL TRIAL: NCT00402909
Title: A 16-week, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Compare the Safety and Efficacy of Nateglinide vs. Placebo in Patients With Type 2 Diabetes Who Are Inadequately Controlled With Basal Insulin Glargine in Combination With Metformin and/or Thiazolidinedione (Pioglitazone or Rosiglitazone)
Brief Title: Safety and Efficacy of Nateglinide in Patients With Type 2 Diabetes Already Taking Insulin Glargine, Metformin and/or Pioglitazone or Rosiglitazone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDJN608AUS13
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes,; fasting glucose,; postprandial glucose,; blood sugar,; HbA1c,; insulin,; glargine,; metformin,; thiazolidinedione
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Nateglinide

INTERVENTIONS:
Drug: Nateglinide

SUMMARY:
This study will assess the safety and efficacy of adding nateglinide to treatment with basal insulin glargine, metformin and/or thiazolidinedione (pioglitazone or rosiglitazone), for patients with type 2 diabetes who are not achieving glycemic control with glargine, metformin and/or thiazolidinedione only.

ELIGIBILITY:
Inclusion Criteria:

* Male/female, age 18-78 inclusive
* Type 2 diabetes, taking glargine, metformin and/or thiazolidinedione for 3 months prior to screening, stable doses for 2 months prior to screening
* HbA1c 7.0-8.5% inclusive
* Fasting plasma glucose <240 mg/dL at screening
* Body Mass Index 22-41 kg/m2

Exclusion Criteria:

* Pregnant or nursing
* Other investigational drugs within 30 days of screening
* Treatment with other anti-diabetic medications other than metformin, glargine and/or thiazolidinedione
* History of type 1 diabetes
* Abnormal kidney function
* History of acute diabetic complications
* Congestive heart failure requiring treatment
* Myocardial infarction, coronary artery surgery, stroke within 6 months of screening
* Liver disease, liver enzymes more than 3 times upper limit of normal
* Fasting triglycerides >700 mg/dL within past 12 weeks
* Acute infections or other conditions that may affect blood sugar or may interfere with interpretation of study data
* Treatment with corticosteroids
* Blood donation within past 12 weeks

Other protocol-defined inclusion/exclusion criterial may apply.

Ages: 18 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin (Hb)_A1c

SECONDARY OUTCOMES:
Change from baseline in 2-hour postprandial glucose during standardized meal test
Proportion of patients achieving American Diabetes Association ADA goal of HbA1c <7.0%
Proportion of patients achieving reduction in HbA1c of 0.5%

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States